CLINICAL TRIAL: NCT04594577
Title: The Clinical Validation of Fluispotter®, a Novel Automated Body-worn System for Serial Sampling of Venous Dried Blood Spots
Brief Title: Clinical Validation of the Fluispotter System for Serial Sampling of Venous Dried Blood Spots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluisense ApS (Industry)
Collaborators: Dantrials Aps (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Fluispotter-01; EUDAMED CIV-20-10-038466 (Other: Danish Medicines Agency); Journal no. 2020100544 (Other: Danish Medicines Agency); Journal no. H-20068538 (Other: Scientific Ethics Committee for the Capital Region, Denmark)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Blood Sampling Procedure; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluispotter (Experimental): Fluispotter automated blood sampling system
  Interventions: Device: Fluispotter

INTERVENTIONS:
Device: Fluispotter — Fluispotter automated blood sampling system applied for venous blood sampling of 20 10 μL samples in a 20 hours sampling session.
  Other Names: Fluispotter Control System, Fluispotter Cartridge, Fluispotter Catheter 45

SUMMARY:
This is a prospective, single-centre, non-comparative, non-randomized, open label, clinical investigation of the clinical performance and safety of Fluispotter. The main aim is to validate the clinical performance and safety of the body-worn Fluispotter system used for automated extraction, collection and storage of 20 dried venous dried blood spot samples of 10 µl over the course of 20 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18
* Able to understand verbal and written instructions in Danish
* Able and willing to sign and date the informed written consent form and letter of authority

Exclusion Criteria:

* Currently participating in a clinical trial evaluating drugs or medical devices
* Known history of coagulation disorders
* Currently taking regular medication (contraceptives, hormonal replacement therapy and antihistamines exempted)
* Regular smoking or use of nicotine products
* Pregnancy
* Haematocrit < 38% (male); < 33% (female)
* Haematocrit > 52% (male); > 48% (female)
* C-reactive protein (CRP) > 10 mg/dL
* Body Mass Index (BMI) > 30
* Known allergies or hypersensitivity to flushing solution constituents
* Other factors which in the opinion of the investigator would interfere with the ability to provide informed consent, comply with study procedures/instructions, or possibly confound the interpretation of the study results or put the subject at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Number of samplings | 20 hours
  Number of successful samplings over a 20-hour period

SECONDARY OUTCOMES:
Clinical safety, safety reporting | 8 ± 2 days
  Frequency and severity of adverse events (AEs), adverse device effects (ADEs) and device deficiencies
Clinical safety, systemic effects | 24 hours
  Clinical haematology and biochemistry tests before and after 20-hour sampling session
Technical performance | 20 hours
  Details of technical performance (yes, no)
Procedure | Approximately 60 minutes and 24 hours
  Details of procedure, including duration of procedure steps (minutes)
Usability: User experience based on questionnaire | 24 hours
  Usability questions related to use and disposal of system (1= Strongly disagree, 2 = Mildly disagree, 3 = Indifferent, 4 = Mildly agree, 5 = Mildly agree)
Usability: Subject experience based on questionnaire | 24 hours and 8 ± 2 days
  Usability questions related to pain and disturbance ((VAS) scale straight horizontal line of fixed length 10 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Sonne, MD, DMSc, Principal Investigator — Dantrials Aps
Locations (1):
- DanTrials ApS, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No